CLINICAL TRIAL: NCT05290844
Title: The Cricoid Force Necessary to Occlude the Esophageal Entrance in Pediatric Patients
Brief Title: The Cricoid Pressure in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procare Riaya Hospital (Other)
Responsible Party: Principal Investigator, Ahed ZEIDAN, Clinical Professor, Procare Riaya Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRH09
Record Dates: First submitted 2022-02-09; First posted 2022-03-22 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Aspiration Pneumonia; Cricoid Cartilage; Pediatric
MeSH Terms: conditions — Pneumonia, Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pediatric cricoid force (Other): one arm ( 3 groups)120 pediatric patients
  Interventions: Other: cricoid pressure

INTERVENTIONS:
Other: cricoid pressure — cricoid force in pediatric patients

SUMMARY:
Because the cricoid force in children has not been quantified, clinicians wrongly used the 'adult' force. it has been found that the use of the adult force can result in compression and distortion of the child's airway and can lead to airway obstruction and difficult intubation. Based on known measurements of the cricoid surface area in children, the theoretical forces necessary to occlude the esophageal entrance have been calculated . These forces were found to be much less than the recommended adult force and much less than the forces that distort the airway as reported previously. Based on these theoretical calculations, the current study was performed to determine the effective cricoid force for pediatric groups (group 1 and group 2).

DETAILED DESCRIPTION:
120 children ASA I or II undergoing different surgeries scheduled to undergo procedures requiring general anesthesia and endotracheal intubation were enrolled in this protocol group1 (40 pts, age 3-5 ysr) group 2 (40 pts,6-8 yrs) and group 3 ( 40 pts, 9-13 yrs) .Following applying of ASA standard monitoring and placement of peripheral iv cannula maximal preoxygenation was achieved (end-tidal oxygen > 90%), and anesthesia was induced with propofol 2 mg/kg, fentanyl 1-1.5 µg/kg and sevoflurane in oxygen/air mixture. Cisatracurium or rocuronuim was given to maintain muscle relaxation. Gentle mask ventilation was begun following an oropharyngeal airway placement. CP was applied by the same anesthesiologist in all patients with his back toward the video monitor. The cricoid cartilage was first identified and then held between the thumb and middle finger and the pressure was applied by the index finger with a force to facilitate the manual ventilation. After loss of consciousness, the force was increased to the predertmined force. The applied cricoid force in successive patients was determined by the response of the previous patient within the same group, using Biased coins up-and-down method in each group. The adjustment force interval was 1 N. Successful insertion of the GT with the adjusted force, was considered ineffective CP and the force was increased 1 N for next patient. Conversely, an unsuccessful GT insertion with the adjusted cricoid force was considered effective CP, and the force was decreased 1 N for the next patient. Tracheal intubation was performed with the appropriate size endotracheal tube while using the same cricoid force, initially tested, and the surgical procedure was begun.

ELIGIBILITY:
Inclusion Criteria:

Age : 3-14 years ASA 1,2 Easy Identification cricoid cartilage No contre indication of CP

Exclusion Criteria:

* ASA 3, 4
* Difficult intubation
* Obese patients
* Contre indication of CP

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
The Cricoid Force Necessary to occlude the Esophageal Entrance In Pediatric patients | day 1
  Measuring the cricoid force using Biased Coin Method ( ED90%) in pediatric patients from 3 years up to 14 years using digital device " the Cricometer "

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Abdulkhaleq, MD, Study Director — PRH
Locations (2):
- Saudi Arabia (2):
  - Procare Riaya Hospital, Khobar, Eastern Province
  - Procare Riaya Hospital, Khobar, Estern

REFERENCES:
- [Derived] Zeidan A, Ramez Salem M, Bamadhaj M, Saifan A, Khorasani A, Mazoit JX, Sadek H, Addelaziz A, Bamadhaj N, Knezevic NN. Quantifying the Effective Cricoid Force to Occlude the Esophageal Entrance in Anesthetized and Muscle-Relaxed Children: A Videolaryngoscopy-Based Assessment. Anaesth Crit Care Pain Med. 2025 Nov 7:101674. doi: 10.1016/j.accpm.2025.101674. Online ahead of print. PMID 41207374